CLINICAL TRIAL: NCT03043196
Title: 1.2% Rosuvastatin Gel As A Local Drug Delivery Agent In Smokers With Chronic Periodontitis- A Randomized Controlled Clinical Trial.
Brief Title: 1.2% Rosuvastatin Gel As A Local Agent In Smokers With Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and HOD, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2014-2015HB
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin Group (Active Comparator): Oral prophylaxis followed by 1.2% Rosuvastatin drug in gel form placed in intrabony defects
  Interventions: Drug: SRP plus Rosuvastatin gel
- Placebo Group (Placebo Comparator): Oral prophylaxis followed by placebo gel placement in intrabony defects
  Interventions: Drug: SRP plus placebo gel

INTERVENTIONS:
Drug: SRP plus Rosuvastatin gel — SRP followed by Rosuvastatin placement into intrabony defect
  Arms: Rosuvastatin Group
Drug: SRP plus placebo gel — SRP followed by placebo gel placement into intrabony defect
  Arms: Placebo Group

SUMMARY:
The purpose of the present study was to evaluate the effects of subgingival delivery of Rosuvastatin gel as an adjunct to scaling and root planing in Smokers With Chronic Periodontitis (CP) patients.

DETAILED DESCRIPTION:
Background: Periodontal diseases are multi-factorial in etiology, and bacteria are one among these etiologic agents. However, mechanical therapy itself may not always reduce or eliminate the anaerobic infection at the base of the pocket, within the gingival tissues. To overcome this, various systemic and local drug delivered antimicrobials have been used as an adjunct to scaling and root planing (SRP).The present study aims to explore the efficacy of 1.2% rosuvastatin (RSV) gel local drug delivery as an adjunct to SRP in smokers with chronic periodontitis (CP).

Methods: Sixty subjects were randomly allocated into two treatment groups: SRP with placebo gel (group 1), SRP with 1.2% RSV gel (group 2). Clinical parameters were recorded at baseline, 6 and 9 months. Radiographic assessment was done using computer aided software at baseline, 6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy CP subjects aged between 30-50 years who are current smokers with no history of periodontal therapy or use of antibiotics in past 6 months, having sites with intrabony defect depth (IBD) ≥ 3mm (distance between alveolar crest and base of the defect on intraoral periapical radiograph) along with PPD ≥5 mm or CAL ≥3 mm in an asymptomatic tooth were included in the study.

A subject was considered as a current smoker if he regularly smoked more than 10 cigarettes/day for a minimum of 5 years

Exclusion Criteria:

* Former smokers, i.e. subjects who had previously been smokers but stopped their habit, and non-smokers were excluded. Subjects allergic to statins, on systemic statin therapy, with any known systemic disease or any other systemic inflammation/ infection which could alter the course of periodontal disease and users of tobacco in any other form than cigarettes were excluded from the study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Defect depth reduction (%) | Change from baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth (mm) | Change from baseline to 9 months
  measured in mm
clinical attachment level (mm) | Change from baseline to 9 months
  measured in mm
modified sulcus bleeding index | Change from baseline to 9 months
  scale from 0-3
Plaque Index | Change from baseline to 9 months
  scale from 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided